CLINICAL TRIAL: NCT04539964
Title: Vagus Nerve Stimulation Using the SetPoint System for Moderate to Severe Rheumatoid Arthritis: The RESET-RA Study
Brief Title: Vagus Nerve Stimulation for Moderate to Severe Rheumatoid Arthritis
Acronym: RESET-RA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SetPoint Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPM-020
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Vagus nerve; vagus nerve stimulating device; drug refractory; permanent implantable; implant
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: An operationally seamless, 2-stage, randomized, double-blind, sham-controlled, multicenter study. Subjects will be assigned randomly in a 1:1 ratio into either a treatment or control group. Subjects assigned to the treatment group will receive active stimulation for 1 min once per day, and those assigned to the control group will receive non-active stimulation for 1 min once per day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, investigators, joint evaluators and study staff will be blinded. Blinding of subjects, joint evaluators and investigators will be assessed at Weeks 4 and 12.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Active stimulation for 1 min once per day
  Interventions: Procedure: Implant Procedure; Drug: Conventional Synthetic DMARD; Device: Active stimulation
- Control (Sham Comparator): Non-active stimulation for 1 min once per day
  Interventions: Procedure: Implant Procedure; Drug: Conventional Synthetic DMARD; Device: Non-active stimulation

INTERVENTIONS:
Procedure: Implant Procedure — The SetPoint System (study device) contains a miniaturized stimulator (implant) that is surgically implanted inside the left side of the neck on the vagus nerve (implant procedure). All eligible subjects will undergo the surgery under general anesthesia in outpatient settings.
  Other Names: Surgical placement of vagus nerve stimulator inside the neck
Drug: Conventional Synthetic DMARD — All subjects will continue to take at least one type of conventional synthetic DMARD at the same stable dose as for 4 weeks prior to consent
  Other Names: Background therapy with conventional synthetic DMARD
Device: Active stimulation — Active stimulation for 1 min once per day
  Arms: Treatment
Device: Non-active stimulation — Non-active stimulation for 1 min once per day
  Arms: Control

SUMMARY:
The RESET-RA study will assess the safety and efficacy of the SetPoint System (study device) for the treatment of adult patients with active, moderate to severe rheumatoid arthritis who have had an inadequate response or intolerance to biologic or targeted synthetic Disease-Modifying Anti-Rheumatic Drugs (DMARDs). The study device contains a miniaturized stimulator (implant) that is surgically placed under general anesthesia on the vagus nerve through a small incision on the left side of the neck (implant procedure). The study will enroll up to 250 subjects at up to 45 sites. All eligible subjects will undergo the implant procedure. Half of the subjects will receive active stimulation (treatment) and the other half will receive non-active stimulation (control). After completing primary endpoint assessments at Week 12, there will be a one-way crossover of control subjects to active stimulation and a 252-week open-label follow-up with all subjects (treatment and control) receiving active stimulation to evaluate long-term safety.

DETAILED DESCRIPTION:
The RESET-RA study is an operationally seamless, 2-stage, randomized, double-blind, sham-controlled, multicenter pivotal study enrolling up to 250 subjects at up to 45 study centers across the U.S. The study will assess the safety and efficacy of the SetPoint System (study device) for the treatment of adult patients with active, moderate to severe rheumatoid arthritis (RA) who have had an inadequate response, loss of response or intolerance to biologic or targeted synthetic Disease-Modifying Anti-Rheumatic Drugs (DMARDs). The study device contains a miniaturized stimulator (implant) that is surgically implanted inside the left side of the neck on the vagus nerve (implant procedure). The implant delivers a small amount of electricity (stimulation) to the nerve. All eligible subjects will undergo the surgery under general anesthesia. Half of the subjects will receive active stimulation (the treatment group) and the other half will receive non-active stimulation (the control group). Stimulation will be delivered for 1 min once per day for 12 weeks. After completing primary endpoint assessments at Week 12, there will be a one-way crossover of control subjects to active stimulation and a 252-week open-label follow-up with all subjects (treatment and control) receiving active stimulation to evaluate long-term safety. Blinding will be maintained until the last enrolled and randomized subject in Stage 2 completes Week 12 assessments, and the study database is locked.

ELIGIBILITY:
Inclusion Criteria:

* 22-75 years of age at screening
* Active moderate or severe RA, defined as at least 4/28 tender and 4/28 swollen joints
* Demonstrated an inadequate response, loss of response, or intolerance to 1 or more approved for rheumatoid arthritis biologic or targeted synthetic Disease-Modifying Anti-Rheumatic Drugs (DMARDs), including Janus kinase inhibitors (JAKi)
* Receiving treatment with at least 1 conventional synthetic DMARD for at least 12 weeks and on a continuous non-changing dose and route of administration for at least 4 weeks prior to Screening and able to continue the same stable dose through Week 12

Exclusion Criteria:

* Untreated or poorly controlled psychiatric illness or history of substance abuse
* Significant immunodeficiency due to underlying illness
* History of stroke or transient ischemic attack, or diagnosis of cerebrovascular fibromuscular dysplasia
* Clinically significant cardiovascular disease
* Neurological syndromes, including multiple sclerosis, Alzheimer's disease, or Parkinson's disease
* Uncontrolled fibromyalgia
* History of left or right carotid surgery
* History of unilateral or bilateral vagotomy, partial or complete splenectomy
* Recurrent vasovagal syncope episodes
* Current, regular use of tobacco products
* Hypersensitivity/allergy to MRI contrast agents and/or unable to perform MRI

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2027-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Tesser, MD, Principal Investigator — Arizona Arthritis and Rheumatology Research, P.C.; Mark Richardson, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (42):
- United States (42):
  - Arizona Arthritis ans Rheumatology Research, PPLC, Mesa, Arizona
  - Arizona Arthritis Rheumatology & Research, PLLC, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Tucson, Arizona
  - Medvin Clinical Research, Covina, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Medvin Clinical Research, Whittier, California
  - The Arthritis & Rheumatology Clinic of Northern Colorado, Fort Collins, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Delaware Arthritis, Lewes, Delaware
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - HARAC Research Corporation, Avon Park, Florida
  - RecioMed Clinical Research Network, Inc., Boynton Beach, Florida
  - Bay Area Rheumatology, Clearwater, Florida
  - IRIS Research and Development, Plantation, Florida
  - Augusta University, Augusta, Georgia
  - Parris and Associates Rheumatology, Lawrenceville, Georgia
  - Northwestern University, Chicago, Illinois
  - Willow Rheumatology and Wellness PLLC, Willowbrook, Illinois
  - Massachusetts General Hospital Division of Rheumatology, Allergy, and Immunology, Boston, Massachusetts
  - June DO, PC, Lansing, Michigan
  - Saint Paul Rheumatology, P.A., Eagan, Minnesota
  - Kansas City Physician Partners, Kansas City, Missouri
  - West County Rheumatology, St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Long Island Regional Arthritis & Osteoporosis Care, Babylon, New York
  - Arthritis & Osteoporosis Consultants Of The Carolinas, Charleston, North Carolina
  - DJL Clinical Research, Charlotte, North Carolina
  - Health Research of Oklahoma, PLLC, Oklahoma City, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Arthritis & Rheumatology Research Institute, PLLC, Allen, Texas
  - Austin Regional Clinic, Austin, Texas
  - Tekton Research, Austin, Texas
  - Central Texas Rheumatology Associates, Austin, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Biopharma Informatic, Houston, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Annapolis Rheumatology, Fairfax, Virginia
  - Sound Clinical Research, LLC, Bothell, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
No sharing data is planned.

REFERENCES:
- [Derived] Tesser JRP, Crowley AR, Box EJ, June JP, Wickersham PB, Valenzuela GJ, Gaylis NB, Lam GKW, Pacheco LA, Ridley DJ, Pinto-Patarroyo GP, Novack SN, Churchill MA, Kohler M, Lee EC, Pando JA, Parris GR, Peterson JR, Shah T, Singhal AK, Vuong V, Levine YA, Evangelista ML, Derosier AA, Curtis JR, Richardson RM, Chernoff D. Vagus nerve-mediated neuroimmune modulation for rheumatoid arthritis: a pivotal randomized controlled trial. Nat Med. 2025 Dec 22. doi: 10.1038/s41591-025-04114-7. Online ahead of print. PMID 41429981
- [Derived] Peterson D, Van Poppel M, Boling W, Santos P, Schwalb J, Eisenberg H, Mehta A, Spader H, Botros J, Vrionis FD, Ko A, Adelson PD, Lega B, Konrad P, Calle G, Vale FL, Bucholz R, Richardson RM. Clinical safety and feasibility of a novel implantable neuroimmune modulation device for the treatment of rheumatoid arthritis: initial results from the randomized, double-blind, sham-controlled RESET-RA study. Bioelectron Med. 2024 Mar 13;10(1):8. doi: 10.1186/s42234-023-00138-x. PMID 38475923

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 405 subjects were consented, and 162 subjects were screen failures. Of the 243 subjects meeting eligibility, 1 subject did not complete the implant procedure per Sponsor decision; the remaining 242 subjects were implanted and subsequently randomly assigned to either treatment with active stimulation (n=122) or control with sham, non-active stimulation (n=120).
Period: Overall Study
Arm/Group | Treatment | Control
Started | 122 | 120
Week 12 (primary endpoint) | 122 (1/122 subjects missed this visit and was imputed as a non-responder) | 120 (1/120 subjects missed this visit and was imputed as a non-responder)
Week 24 | 119 (1/122 subjects discontinued, 2/122 subjects missed this visit) | 117 (3/120 subjects missed this visit)
Week 36 | 119 (2/122 subjects discontinued, 1/122 subjects missed this visit) | 115 (1/120 subjects discontinued, 4/120 subjects missed this visit)
Week 48 | 119 (2/122 subjects discontinued, 1/122 subjects missed this visit) | 114 (4/120 subjects discontinued, 2/120 subjects missed this visit)
Completed | 120 | 116
Not Completed | 2 | 4
Not completed — device malfunction | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Active stimulation for 1 min once per day
  Implant Procedure: The SetPoint System (study device) contains a miniaturized stimulator (implant) that is surgically implanted inside the left side of the neck on the vagus nerve (implant procedure). All eligible subjects will undergo the surgery under general anesthesia in outpatient settings.
  Conventional Synthetic Disease-Modifying Antirheumatic Drug (DMARD): All subjects will continue to take at least one type of conventional synthetic DMARD at the same stable dose as for 4 weeks prior to consent
  Active stimulation: Active stimulation for 1 minute once per day
- Control: Non-active stimulation for 1 min once per day
  Implant Procedure: The SetPoint System (study device) contains a miniaturized stimulator (implant) that is surgically implanted inside the left side of the neck on the vagus nerve (implant procedure). All eligible subjects will undergo the surgery under general anesthesia in outpatient settings.
  Conventional Synthetic DMARD: All subjects will continue to take at least one type of conventional synthetic DMARD at the same stable dose as for 4 weeks prior to consent
  Non-active stimulation: Non-active stimulation for 1 minute once per day
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 122 | 120 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (10.28) | 55.5 (10.49) | 55.7 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 110 | 208
  Male | 24 | 10 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 22 | 45
  Not Hispanic or Latino | 98 | 95 | 193
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 12 | 22
  White | 102 | 93 | 195
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 122 | 120 | 242
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.7 (7.25) | 29.8 (6.71) | 30.3 (6.98)
Rheumatoid arthritis (RA) duration [Mean (Standard Deviation); unit: years] | 13.0 (10.59) | 11.8 (10.45) | 12.4 (10.52)
Clinical Disease Activity Index (CDAI) score [Mean (Standard Deviation); unit: score on a scale] | 36.1 (12.60) | 38.2 (12.75) | 37.1 (12.69)
Disease Activity Score-28 with C-reactive protein (DAS28-CRP) score [Mean (Standard Deviation); unit: score on a scale] | 5.3 (0.91) | 5.4 (0.96) | 5.3 (0.93)
Rheumatoid Factor (RF) [Count of Participants; unit: Participants]
  Negative | 73 | 64 | 137
  Positive | 49 | 56 | 105
Anti-Citrullinated Protein Antibodies (ACPA) [Count of Participants; unit: Participants]
  Negative | 57 | 61 | 118
  Positive | 61 | 59 | 120
  Missing | 4 | 0 | 4
Serology [Count of Participants; unit: Participants]
  Negative | 56 | 54 | 110
  Positive | 62 | 66 | 128
  Missing | 4 | 0 | 4
Prior b/tsDMARDs [Mean (Standard Deviation); unit: number of b/tsDMARDs] | 2.5 (1.98) | 2.7 (1.87) | 2.6 (1.92)
Number of prior b/tsDMARDs [Count of Participants; unit: Participants]
  1 | 52 | 42 | 94
  2 | 25 | 28 | 53
  3 | 15 | 16 | 31
  4 | 15 | 15 | 30
  5 | 7 | 8 | 15
  6 | 2 | 5 | 7
  7 | 2 | 4 | 6
  8 | 2 | 1 | 3
  9 | 0 | 0 | 0
  10+ | 2 | 1 | 3
Tender Joint Count (out of 28 joints) [Mean (Standard Deviation); unit: number of joints] | 14.1 (6.94) | 15.0 (7.26) | 14.6 (7.10)
Swollen Joint Count (out of 28 joints) [Mean (Standard Deviation); unit: number of joints] | 9.6 (5.46) | 10.5 (4.98) | 10.0 (5.23)
HAQ-DI Score [Mean (Standard Deviation); unit: score on a scale] | 1.4 (0.59) | 1.3 (0.61) | 1.4 (0.60)
Pain (0-10) [Mean (Standard Deviation); unit: score on a scale] | 5.5 (2.00) | 5.7 (2.23) | 5.6 (2.12)
Subject's Global Assessment (0-10) [Mean (Standard Deviation); unit: score on a scale] | 6.2 (2.07) | 6.0 (2.25) | 6.1 (2.16)
Evaluator's Global Assessment (0-10) [Mean (Standard Deviation); unit: score on a scale] | 6.3 (1.88) | 6.7 (1.72) | 6.5 (1.80)
hsCRP [Mean (Standard Deviation); unit: mg/L] | 8.41 (12.338) | 8.01 (12.762) | 8.21 (12.526)

OUTCOME MEASURES:

1. Primary Outcome: the American College of Rheumatology (ACR) 20 Response
Description: Response is defined as achieving at least 20% improvement from baseline to Week 12 in tender and swollen joint counts of 28 joints (scale 0=best to 28=worst) and 3 out of the following 5 measures: Health Assessment Questionnaire Disability Index (HAQ-DI) score (scale 0=no difficulty to 3=unable to do), subject global assessment (0=best to 10=worst), subject pain (0=no pain to 10=worst), evaluator's global assessment (0=best to 10=worst), or high sensitivity C-reactive protein (hsCRP) concentration (mg/L).
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 122 | 120
Participants | 43 | 29
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — The null hypothesis (H0) is that there is no difference between the treatment and control groups versus the alternative hypothesis (H1) that treatment group response rate exceeds the control group response rate; p = 0.0209, Cochran-Mantel-Haenszel — The study is considered successful if there is a statistically significant improvement in the proportion of subjects with ACR20 response in favor of the SetPoint System at the one-sided alpha of 0.025; Risk Difference (RD) = 11.8, 95% CI 2-sided [0.6 to 23.1]

2. Secondary Outcome: DAS28-CRP Good or Moderate Response as Defined by European League Against Rheumatism (EULAR)
Description: The Disease Activity Score in 28 joints calculated with C-reactive protein (DAS28-CRP) good or moderate response as defined by EULAR based on a composite score of 4 items: tender and swollen joint counts of 28 joints (scale 0=best to 28=worst), subject global assessment (0=best to 10=worst) and high-sensitivity C-reactive protein (hsCRP) concentration (mg/L). A total score ranges from 0 to 10 and is computed as follows:
  DAS28-CRP = 0.56 * sqrt(TJC28) + 0.28 * sqrt(SJC28) + 0.36 * ln(CRP+1) + 0.014 * SGA + 0.96
  A subject is considered having a moderate treatment response if:
  * DAS28-CRP score improvement from baseline to Week 12 is > 0.6 and ≤ 1.2, and the DAS28-CRP score at Week 12 is ≤ 5.1; or
  * DAS28-CRP score improvement from baseline to Week 12 is > 1.2, and the DAS28-CRP score at Week 12 is > 3.2.
  A subject is considered having a good treatment response if:
  • DAS28-CRP score improvement from baseline to Week 12 is > 1.2 and the DAS28-CRP score at Week 12 is ≤ 3.2
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 122 | 120
Participants | 74 | 50
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0048, Cochran-Mantel-Haenszel — Adjusted p-value. Hochberg's step-up procedure was used to control the family wise type 1 error rate at a 1-sided significance level of 0.025; Risk Difference (RD) = 19.5, 95% CI 2-sided [7.3 to 31.7]

3. Secondary Outcome: DAS28-CRP Response (MCID -1.2) at Week 12
Description: The Disease Activity Score in 28 joints calculated with C-reactive protein (DAS28-CRP) response is based on the minimal clinically important difference (MCID) of -1.2 from baseline.
  DAS28-CRP is based on a composite score of 4 items: tender and swollen joint counts of 28 joints (scale 0=best to 28=worst), subject global assessment (0=best to 10=worst) and high-sensitivity C-reactive protein (hsCRP) concentration (mg/L). A total score ranges from 0 to 10 and is computed as follows:
  DAS28-CRP = 0.56 * sqrt(TJC28) + 0.28 * sqrt(SJC28) + 0.36 * ln(CRP+1) + 0.014 * SGA + 0.96
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 122 | 120
Participants | 55 | 39
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0528, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 13.2, 95% CI 2-sided [1.1 to 25.3]

4. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Response (MCID -0.22)
Description: HAQ-DI response based on the MCID of -0.22 from baseline.
  The HAQ-DI is a questionnaire validated for RA self-assessment by subjects that contains 20 questions in the following 8 functional areas:
  * Dressing and grooming
  * Arising
  * Eating
  * Walking
  * Hygiene
  * Reach
  * Grip
  * Common daily activities
  Scoring within each functional area is from 0 (without any difficulty) to 3 (unable to do). The total score is obtained by summing 8 area scores and dividing by 8. The total HAQ-DI score ranges from 0 to 3 and corresponds to the current degree of disability:
  * 0 to < 1 Mild difficulties to moderate disability
  * 1 to < 2 Moderate disability
  * 2 to 3 Severe to very severe disability
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 122 | 120
Participants | 56 | 44
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0797, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 9.0, 95% CI 2-sided [-3.3 to 21.4]

5. Secondary Outcome: ACR20 Response at Week 12 From Day 0
Description: Response is defined as achieving at least 20% improvement from Day 0 to Week 12 in tender and swollen joint counts of 28 joints (scale 0=best to 28=worst) and 3 out of the following 5 measures: Health Assessment Questionnaire Disability Index (HAQ-DI) score (scale 0=no difficulty to 3=unable to do), subject global assessment (0=best to 10=worse), subject pain (0=no pain to 10=worst), evaluator's global assessment (0=best to 10=worst), or high sensitivity C-reactive protein (hsCRP) concentration (mg/mL).
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 122 | 120
Participants | 38 | 27
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0797, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 8.0, 95% CI 2-sided [-3.1 to 19.0]

6. Other Pre Specified Outcome: Bone Erosion Progression, All Completers
Description: RAMRIS is a standardized system for RA MRI scoring of 4 different types of joint pathologies in the wrist and the hand. A total score for each pathology is generated by the summation of individual joint/bone scores as follows:
  * Synovitis: 8 joints each scored on a scale from 0 = normal to 3 = severe, resulting in a total score from 0 to 24.
  * Bone erosion: 25 bones each scored on a scale from 0 (0-10% eroded volume) to 10 (91-100% eroded volume), resulting in a total score from 0 to 250.
  * Osteitis: 25 bones scored on a scale from 0 (no osteitis) to 3 (68-100% of bone volume involved), resulting in a total score from 0 to 75.
  * CARLOS (cartilage loss): 25 joints each scored on a scale from 0 (no damage) to 4 (complete ankylosis or fusion), resulting in a total score from 0 to 100.
  The proportion of bone erosion progressors is the % subjects with an increase of > 0.5 on the bone erosion score, comparing baseline to Week 12. An increase of > 0.5 represents disease progression.
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 108 | 105
Participants | 18 | 21
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — The null hypothesis (H0) is that there is no difference between the treatment and control groups versus the alternative hypothesis (H1) that control group response rate exceeds the treatment group response rate; p = 0.2476, Cochran-Mantel-Haenszel; Risk Difference (RD) = -3.7, 95% CI 2-sided [-14.4 to 7.0]

7. Other Pre Specified Outcome: Bone Erosion Progression, All Completers With Erosive Phenotype
Description: as for outcome 6
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Count of Participants; unit: Participants
Groups:
- Treatment, Erosive Phenotype: Subgroup of subjects receiving active stimulation for 1 min once per day that have an erosive phenotype. Subjects meeting the subgroup criteria for having an erosive phenotype had a baseline synovitis score of 2 or more on any joint; or, if none of the joints score greater than 2, had at least 4 joints with a score of 1 at baseline; or had any joint with osteitis (score of 1 or more) at baseline.
- Control, Erosive Phenotype: Subgroup of subjects receiving non-active stimulation for 1 min once per day that have an erosive phenotype. Subjects meeting the subgroup criteria for having an erosive phenotype had a baseline synovitis score of 2 or more on any joint; or, if none of the joints score greater than 2, had at least 4 joints with a score of 1 at baseline; or had any joint with osteitis (score of 1 or more) at baseline.
Arm/Group | Treatment, Erosive Phenotype | Control, Erosive Phenotype
Number analyzed (Participants) | 53 | 45
Participants | 10 | 17
Statistical Analysis 1: Comparison: Treatment, Erosive Phenotype vs Control, Erosive Phenotype; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.0156, Cochran-Mantel-Haenszel; Risk Difference (RD) = -20.2, 95% CI 2-sided [-38.1 to -2.2]

8. Other Pre Specified Outcome: Bone Erosion Progression, All Completers That Previously Only Failed 1 b/tsDMARD
Description: as for outcome 6
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Count of Participants; unit: Participants
Groups:
- Treatment, 1 Prior b/tsDMARD: Subgroup of subjects receiving active stimulation for 1 min once per day that have previously only failed 1 b/tsDMARD
- Control, 1 Prior b/tsDMARD: Subgroup of subjects receiving non-active stimulation for 1 min once per day that have previously only failed 1 b/tsDMARD
Arm/Group | Treatment, 1 Prior b/tsDMARD | Control, 1 Prior b/tsDMARD
Number analyzed (Participants) | 46 | 36
Participants | 3 | 9
Statistical Analysis 1: Comparison: Treatment, 1 Prior b/tsDMARD vs Control, 1 Prior b/tsDMARD; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.0099, Cochran-Mantel-Haenszel; Risk Difference (RD) = -18.6, 95% CI 2-sided [-34.7 to -2.6]

9. Other Pre Specified Outcome: Change in Erosion Score, All Completers
Description: RAMRIS is a standardized system for RA MRI scoring of 4 different types of joint pathologies in the wrist and the hand (synovitis, bone erosion, osteitis, and cartilage loss). A total score for each pathology is generated by the summation of individual joint/bone scores:
  • Bone erosion: 25 bones each scored on a scale from 0 (0-10% eroded volume) to 10 (91-100% eroded volume), resulting in a total score from 0 to 250.
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 108 | 105
score on a scale | 0.2 (0.85) | 0.5 (1.74)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — The null hypothesis (H0) is that there is no difference between the treatment and control groups versus the alternative hypothesis (H1) that the control group mean change exceeds the treatment group mean change; p = 0.0618, Mixed Models Analysis; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.8 to 0.1]

10. Other Pre Specified Outcome: Change in Erosion Score, All Completers With Erosive Phenotype
Description: as for outcome 9
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment, Erosive Phenotype | Control, Erosive Phenotype
Number analyzed (Participants) | 53 | 45
score on a scale | 0.3 (1.09) | 1.1 (2.51)
Statistical Analysis 1: Comparison: Treatment, Erosive Phenotype vs Control, Erosive Phenotype; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.0308, Mixed Models Analysis; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.8 to 0.0]

11. Other Pre Specified Outcome: Change in Erosion Score, All Completers That Previously Only Failed 1 b/tsDMARD
Description: as for outcome 9
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment, 1 Prior b/tsDMARD | Control, 1 Prior b/tsDMARD
Number analyzed (Participants) | 46 | 36
score on a scale | 0.0 (0.60) | 0.8 (2.57)
Statistical Analysis 1: Comparison: Treatment, 1 Prior b/tsDMARD vs Control, 1 Prior b/tsDMARD; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.0441, Mixed Models Analysis; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.7 to 0.1]

12. Other Pre Specified Outcome: Change in Synovitis Score, All Completers
Description: RAMRIS is a standardized system for RA MRI scoring of 4 different types of joint pathologies in the wrist and the hand (synovitis, bone erosion, osteitis, and cartilage loss). A total score for each pathology is generated by the summation of individual joint/bone scores:
  • Synovitis: 8 joints each scored on a scale from 0 = normal to 3 = severe, resulting in a total score from 0 to 24.
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 108 | 105
score on a scale | 0.0 (1.64) | 0.1 (1.51)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.2871, Mixed Models Analysis; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.6 to 0.3]

13. Other Pre Specified Outcome: Change in Synovitis Score, All Completers With Erosive Phenotype
Description: as for outcome 12
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment, Erosive Phenotype | Control, Erosive Phenotype
Number analyzed (Participants) | 53 | 45
score on a scale | -0.1 (2.27) | 0.0 (1.77)
Statistical Analysis 1: Comparison: Treatment, Erosive Phenotype vs Control, Erosive Phenotype; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.4345, Mixed Models Analysis; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.9 to 0.7]

14. Other Pre Specified Outcome: Change in Synovitis Score, All Completers That Previously Only Failed 1 b/tsDMARD
Description: as for outcome 12
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment, 1 Prior b/tsDMARD | Control, 1 Prior b/tsDMARD
Number analyzed (Participants) | 46 | 36
score on a scale | 0.1 (0.81) | 0.6 (1.78)
Statistical Analysis 1: Comparison: Treatment, 1 Prior b/tsDMARD vs Control, 1 Prior b/tsDMARD; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.0900, Mixed Models Analysis; Mean Difference (Net) = -0.45, 95% CI 2-sided [-1.1 to 0.2]

15. Other Pre Specified Outcome: Change in Osteitis Score, All Completers
Description: RAMRIS is a standardized system for RA MRI scoring of 4 different types of joint pathologies in the wrist and the hand (synovitis, bone erosion, osteitis, and cartilage loss). A total score for each pathology is generated by the summation of individual joint/bone scores:
  • Osteitis: 25 bones scored on a scale from 0 (no osteitis) to 3 (68-100% of bone volume involved), resulting in a total score from 0 to 75.
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 108 | 104
score on a scale | 0.1 (2.61) | 0.8 (4.13)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.0662, Mixed Models Analysis; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.7 to 0.2]

16. Other Pre Specified Outcome: Change in Osteitis Score, All Completers With Erosive Phenotype
Description: as for outcome 15
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment, Erosive Phenotype | Control, Erosive Phenotype
Number analyzed (Participants) | 53 | 45
score on a scale | 0.2 (3.74) | 1.8 (6.18)
Statistical Analysis 1: Comparison: Treatment, Erosive Phenotype; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.0450, Mixed Models Analysis; Mean Difference (Net) = -1.8, 95% CI 2-sided [-3.9 to 0.3]

17. Other Pre Specified Outcome: Change in Osteitis Score, All Completers That Previously Only Failed 1 b/tsDMARD
Description: as for outcome 15
Time Frame: Week 12
Population: ITT with MRI images at both Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment, 1 Prior b/tsDMARD | Control, 1 Prior b/tsDMARD
Number analyzed (Participants) | 46 | 36
score on a scale | -0.3 (2.22) | 1.1 (4.92)
Statistical Analysis 1: Comparison: Treatment, 1 Prior b/tsDMARD vs Control, 1 Prior b/tsDMARD; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.0350, Mixed Models Analysis; Mean Difference (Net) = -1.55, 95% CI 2-sided [-3.2 to 0.1]

18. Other Pre Specified Outcome: Clinical Disease Activity Index (CDAI) Low Disease Activity (LDA) or Remission
Description: The CDAI score is based on 4 items:
  * TJC28, tender joint count of 28 joints (scale 0=best to 28=worst)
  * SJC28, swollen joint count of 28 joints (scale 0=best to 28=worst)
  * SGA, subject global assessment (0=best to 10=worst)
  * EGA, evaluator's global assessment (0=best to 10=worst)
  The CDAI score is calculated as follows and ranges from 0 to 76:
  • CDAI = TJC28 + SJC28 + SGA + EGA
  The CDAI score corresponds to the current RA activity:
  * 0 to ≤ 2.8 Remission
  * >2.8 to ≤ 10 Low disease activity (LDA)
  * >10 to ≤ 22 Moderate disease activity
  * > 22 High disease activity
Time Frame: Week 12
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 120 | 119
Participants | 28 | 19
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0648, Cochran-Mantel-Haenszel; Risk Difference (RD) = 7.8, 95% CI 2-sided [-2.1 to 17.7]

19. Other Pre Specified Outcome: DAS28-CRP Low Disease Activity (LDA) or Remission
Description: The Disease Activity Score in 28 joints calculated with C-reactive protein (DAS28-CRP) score is a composite index providing a measure of disease activity, comprising:
  * TJC28, tender joint count of 28 joints (scale 0=best to 28=worst)
  * SJC28, swollen joint count of 28 joints (scale 0=best to 28=worst)
  * SGA, subject global assessment (0=best to 10=worst)
  * hsCRP (mg/L), high sensitivity C-reactive protein concentration (mg/L)
  A total score ranges from 0 to 10 and is computed as follows:
  DAS28-CRP = 0.56 * sqrt(TJC28) + 0.28 * sqrt(SJC28) + 0.36 * ln(CRP+1) + 0.014 * SGA + 0.96
  The DAS28-CRP score corresponds to the current RA activity:
  * 0 to < 2.6 Remission
  * 2.6 to < 3.2 LDA
  * 3.2 to ≤ 5.1 Moderate activity
  * > 5.1 High activity
Time Frame: Week 12
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 119 | 119
Participants | 31 | 18
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0154, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.4, 95% CI 2-sided [1.2 to 21.6]

20. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, All Completers
Description: as for outcome 1
Time Frame: Week 24
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Groups:
- Treatment to Open Label (TOL): Treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- Control to Open Label (COL): Control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- All (TOL+COL): Combination of TOL and COL populations
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 117 | 236
Participants | 53 | 65 | 118

21. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, Non-augmented
Description: as for outcome 1
Time Frame: Week 24
Population: Subgroup of subjects receiving active stimulation for 1 min once per day, whose study therapy has not been augmented, who completed assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment to Open Label (TOL), Non-augmented: A subgroup of subjects from the TOL population who did not have study therapy augmented during the outcome measure timeframe.
  Augmentation of study therapy means the addition of treatment for RA therapy to active stimulation applied after completion of Week 12 assessments, during open-label, long-term follow-up. Augmented therapy may be applied at any time during long-term follow-up. The decision about the need, type and timing of treatment is left to the discretion of the Co-PI Rheumatologist and the subject. Subjects combining active stimulation with the following additions to RA therapy fall into the augmented therapy subgroup for analysis of response rates for key efficacy endpoints at specific timepoints:
  * Prednisone equivalent >10 mg/day. If average daily corticosteroid use exceeds 10 mg/day prednisone after a period (time from previous visit up to the day before the current visit), the subject is assigned to the augmented therapy subgroup for that visit.
  * Corticosteroid injection. If subject received a corticosteroid injection within 30 days prior to a study visit, the subject is assigned to the augmented therapy subgroup for that visit.
  * b/ts/csDMARD. Subjects who receive treatment with biologic, targeted synthetic, or additional conventional synthetic DMARD, or increased dose of background conventional synthetic DMARD will be assigned to the augmented therapy subgroup for all subsequent visits.
- Control to Open Label (COL), Non-augmented: A subgroup of subjects from the COL population who did not have study therapy augmented during the outcome measure timeframe.
  Augmentation of study therapy means the addition of treatment for RA therapy to active stimulation applied after completion of Week 12 assessments, during open-label, long-term follow-up. Augmented therapy may be applied at any time during long-term follow-up. The decision about the need, type and timing of treatment is left to the discretion of the Co-PI Rheumatologist and the subject. Subjects combining active stimulation with the following additions to RA therapy fall into the augmented therapy subgroup for analysis of response rates for key efficacy endpoints at specific timepoints:
  * Prednisone equivalent >10 mg/day. If average daily corticosteroid use exceeds 10 mg/day prednisone after a period (time from previous visit up to the day before the current visit), the subject is assigned to the augmented therapy subgroup for that visit.
  * Corticosteroid injection. If subject received a corticosteroid injection within 30 days prior to a study visit, the subject is assigned to the augmented therapy subgroup for that visit.
  * b/ts/csDMARD. Subjects who receive treatment with biologic, targeted synthetic, or additional conventional synthetic DMARD, or increased dose of background conventional synthetic DMARD will be assigned to the augmented therapy subgroup for all subsequent visits.
- All (TOL Non-augmented+COL Non Augmented): Combination of the non-augmented TOL and COL populations
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 96 | 98 | 194
Participants | 50 | 52 | 102

22. Other Pre Specified Outcome: Clinical Disease Activity Index (CDAI) Low Disease Activity (LDA) or Remission, All Completers
Description: as for outcome 18
Time Frame: Week 24
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 117 | 236
Participants | 33 | 36 | 69

23. Other Pre Specified Outcome: Clinical Disease Activity Index (CDAI) Low Disease Activity (LDA) or Remission, Non-augmented
Description: as for outcome 18
Time Frame: Week 24
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 96 | 98 | 194
Participants | 33 | 31 | 64

24. Other Pre Specified Outcome: DAS28-CRP Low Disease Activity (LDA) or Remission, All Completers
Description: as for outcome 19
Time Frame: Week 24
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 118 | 117 | 235
Participants | 36 | 37 | 73

25. Other Pre Specified Outcome: DAS28-CRP Low Disease Activity (LDA) or Remission, Non-augmented
Description: as for outcome 19
Time Frame: Week 24
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 95 | 98 | 193
Participants | 35 | 32 | 67

26. Other Pre Specified Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) MCID Response, All Completers
Description: as for outcome 4
Time Frame: Week 24
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 117 | 236
Participants | 64 | 72 | 136

27. Other Pre Specified Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Response (MCID -0.22), Non-augmented
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 96 | 98 | 194
Participants | 56 | 62 | 118

28. Other Pre Specified Outcome: Study Participants That Are Somewhat to Very Satisfied With the SetPoint System for Treatment of Rheumatoid Arthritis
Description: Patient satisfaction was assessed at Week 24 using five-point Likert rating scale:
  * I am very dissatisfied
  * I am somewhat dissatisfied
  * I am neither satisfied nor dissatisfied
  * I am somewhat satisfied
  * I am very satisfied
Time Frame: Week 24
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 114 | 233
Participants | 90 | 92 | 182

29. Other Pre Specified Outcome: Study Participants That Are Neither Satisfied Nor Dissatisfied With the SetPoint System for Treatment of Rheumatoid Arthritis
Description: as for outcome 28
Time Frame: Week 24
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 114 | 233
Participants | 14 | 12 | 26

30. Other Pre Specified Outcome: Study Participants That Are Somewhat to Very Dissatisfied With the SetPoint System for Treatment of Rheumatoid Arthritis
Description: as for outcome 28
Time Frame: Week 24
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 114 | 233
Participants | 15 | 10 | 25

31. Other Pre Specified Outcome: Study Participants That Would Recommend the SetPoint System to a Family Member or Friend
Description: Patients were asked a question about whether they would recommend the SetPoint System to family and friends
Time Frame: Week 24
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 118 | 114 | 232
Participants | 108 | 110 | 218

32. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, All Completers
Description: as for outcome 1
Time Frame: Week 36
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 115 | 234
Participants | 57 | 64 | 121

33. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, Non-augmented
Description: as for outcome 1
Time Frame: Week 36
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 89 | 87 | 176
Participants | 46 | 54 | 100

34. Other Pre Specified Outcome: Clinical Disease Activity Index (CDAI) Low Disease Activity (LDA) or Remission, All Completers
Description: as for outcome 18
Time Frame: Week 36
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 117 | 114 | 231
Participants | 39 | 40 | 79

35. Other Pre Specified Outcome: Clinical Disease Activity Index (CDAI) Low Disease Activity (LDA) or Remission, Non-augmented
Description: as for outcome 18
Time Frame: Week 36
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 87 | 87 | 174
Participants | 34 | 35 | 69

36. Post Hoc Outcome: Persistence With SetPoint System as a Stand-alone Therapy
Description: Therapy persistence means continuation of therapy after it is initiated.
Time Frame: Week 24
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 96 | 99 | 195

37. Post Hoc Outcome: Persistence With SetPoint System Therapy Augmented With a b/tsDMARD
Description: Therapy persistence means the continuation of therapy after it is initiated.
  Augmentation of study therapy means the addition of treatment for RA therapy to active stimulation applied after completion of Week 12 assessments, during open-label, long-term follow-up. Augmented therapy may be applied at any time during long-term follow-up. The decision about the need, type and timing of treatment is left to the discretion of the Co-PI Rheumatologist and the subject. Subjects combining active stimulation with the following additions to RA therapy fall into the augmented therapy subgroup for analysis of response rates for key efficacy endpoints at specific timepoints:
  * Prednisone equivalent >10 mg/day. If average daily corticosteroid use exceeds 10 mg/day prednisone after a period (time from previous visit up to the day before the current visit), the subject is assigned to the augmented therapy subgroup for that visit.
  * Corticosteroid injection. If subject received a corti
Time Frame: Week 24
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 17 | 12 | 29

38. Post Hoc Outcome: Persistence With SetPoint System Therapy Augmented With a csDMARD and/or Steroid
Description: Therapy persistence means continuation of therapy after it is initiated.
  Augmentation of study therapy means the addition of treatment for RA therapy to active stimulation applied after completion of Week 12 assessments, during open-label, long-term follow-up. Augmented therapy may be applied at any time during long-term follow-up. The decision about the need, type and timing of treatment is left to the discretion of the Co-PI Rheumatologist and the subject. Subjects combining active stimulation with the following additions to RA therapy fall into the augmented therapy subgroup for analysis of response rates for key efficacy endpoints at specific timepoints:
  * Prednisone equivalent >10 mg/day. If average daily corticosteroid use exceeds 10 mg/day prednisone after a period (time from previous visit up to the day before the current visit), the subject is assigned to the augmented therapy subgroup for that visit.
  * Corticosteroid injection. If subject received a corticosteroi
Time Frame: Week 24
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 9 | 8 | 17

39. Post Hoc Outcome: Persistence With SetPoint System Therapy as a Stand-alone or Augmented Thereapy
Description: Therapy persistence is defined as the continuation of therapy after it is initiated.
Time Frame: Week 24
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 120 | 118 | 238

40. Post Hoc Outcome: Discontinuation of SetPoint System Therapy
Description: Discontinuation means active stimulation was suspended or the SetPoint System Implant was removed
Time Frame: Week 24
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 2 | 2 | 4

41. Other Pre Specified Outcome: DAS28-CRP Low Disease Activity (LDA) or Remission, All Completers
Description: as for outcome 19
Time Frame: Week 36
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 114 | 107 | 221
Participants | 38 | 40 | 78

42. Other Pre Specified Outcome: DAS28-CRP Low Disease Activity (LDA) or Remission, Non-augmented
Description: as for outcome 19
Time Frame: Week 36
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 85 | 82 | 167
Participants | 31 | 35 | 66

43. Other Pre Specified Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) MCID Response, All Completers
Description: as for outcome 4
Time Frame: Week 36
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 118 | 115 | 233
Participants | 68 | 67 | 135

44. Other Pre Specified Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Response (MCID -0.22), Non-augmented
Description: as for outcome 4
Time Frame: Week 36
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 89 | 87 | 176
Participants | 53 | 51 | 104

45. Post Hoc Outcome: Persistence With SetPoint System as a Stand-alone Therapy
Description: Therapy persistence means continuation of therapy after it is initiated.
Time Frame: Week 36
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 89 | 88 | 177

46. Post Hoc Outcome: Persistence With SetPoint System Therapy Augmented With a b/tsDMARD
Description: as for outcome 37
Time Frame: Week 36
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 25 | 22 | 47

47. Post Hoc Outcome: Persistence With SetPoint System Therapy Augmented With a csDMARD and/or Steroid
Description: as for outcome 38
Time Frame: Week 36
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 7 | 9 | 16

48. Post Hoc Outcome: Persistence With SetPoint System Therapy as a Stand-alone or Augmented Thereapy
Description: Therapy persistence is defined as the continuation of therapy after it is initiated.
Time Frame: Week 36
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 120 | 116 | 236

49. Post Hoc Outcome: Discontinuation of SetPoint System Therapy
Description: Discontinuation means active stimulation was suspended or the SetPoint System Implant was removed
Time Frame: Week 36
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 2 | 4 | 6

50. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, All Completers
Description: as for outcome 1
Time Frame: Week 48
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 114 | 233
Participants | 61 | 62 | 123

51. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, Non-augmented
Description: as for outcome 1
Time Frame: Week 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 77 | 80 | 157
Participants | 43 | 48 | 91

52. Other Pre Specified Outcome: Clinical Disease Activity Index (CDAI) Low Disease Activity (LDA) or Remission, All Completers
Description: as for outcome 18
Time Frame: Week 48
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 118 | 114 | 232
Participants | 47 | 41 | 88

53. Other Pre Specified Outcome: Clinical Disease Activity Index (CDAI) Low Disease Activity (LDA) or Remission, Non-augmented
Description: as for outcome 18
Time Frame: Week 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 76 | 81 | 156
Participants | 36 | 33 | 69

54. Other Pre Specified Outcome: DAS28-CRP Low Disease Activity (LDA) or Remission, All Completers
Description: as for outcome 19
Time Frame: Week 48
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 117 | 111 | 228
Participants | 50 | 42 | 92

55. Other Pre Specified Outcome: DAS28-CRP Low Disease Activity (LDA) or Remission, Non-augmented
Description: as for outcome 19
Time Frame: Week 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 75 | 78 | 153
Participants | 37 | 32 | 69

56. Other Pre Specified Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) MCID Response, All Completers
Description: as for outcome 4
Time Frame: Week 48
Population: ITT, all completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 119 | 113 | 232
Participants | 66 | 67 | 133

57. Other Pre Specified Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Response (MCID -0.22), Non-augmented
Description: as for outcome 4
Time Frame: Week 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL), Non-augmented | Control to Open Label (COL), Non-augmented | All (TOL Non-augmented+COL Non Augmented)
Number analyzed (Participants) | 77 | 80 | 157
Participants | 41 | 49 | 90

58. Post Hoc Outcome: Persistence With SetPoint System as a Stand-alone Therapy
Description: Therapy persistence means continuation of therapy after it is initiated.
Time Frame: Week 48
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 77 | 81 | 158

59. Post Hoc Outcome: Persistence With SetPoint System Therapy Augmented With a b/tsDMARD
Description: as for outcome 37
Time Frame: Week 48
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 32 | 28 | 60

60. Post Hoc Outcome: Persistence With SetPoint System Therapy Augmented With a csDMARD and/or Steroid
Description: as for outcome 38
Time Frame: Week 48
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 16 | 12 | 28

61. Post Hoc Outcome: Persistence With SetPoint System Therapy as a Stand-alone or Augmented Thereapy
Description: Therapy persistence is defined as the continuation of therapy after it is initiated.
Time Frame: Week 48
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 120 | 116 | 236

62. Post Hoc Outcome: Discontinuation of SetPoint System Therapy
Description: Discontinuation means active stimulation was suspended or the SetPoint System Implant was removed
Time Frame: Week 48
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment to Open Label (TOL) | Control to Open Label (COL) | All (TOL+COL)
Number analyzed (Participants) | 122 | 120 | 242
Participants | 2 | 4 | 6

63. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, Subjects With 1 Prior b/tsDMARD
Description: as for outcome 1
Time Frame: Week 12
Population: ITT, subgroup of subjects that previously failed 1 b/tsDMARD
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 52 | 42
Participants | 23 | 8
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0054, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.2, 95% CI 2-sided [7.1 to 43.3]

64. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, Subjects With 2 Prior b/tsDMARD
Description: as for outcome 1
Time Frame: Week 12
Population: ITT, subgroup of subjects that previously failed 2 b/tsDMARD
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 25 | 28
Participants | 8 | 3
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0437, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.3, 95% CI 2-sided [-2.2 to 42.9]

65. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, Subjects With 3 Prior b/tsDMARD
Description: as for outcome 1
Time Frame: Week 12
Population: ITT, subgroup of subjects that previously failed 3 b/tsDMARD
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 16
Participants | 3 | 6
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1643, Cochran-Mantel-Haenszel; Risk Difference (RD) = -17.6, 95% CI 2-sided [-51.1 to 16.0]

66. Other Pre Specified Outcome: the American College of Rheumatology (ACR) 20 Response, Subjects With >=4 Prior b/tsDMARD
Description: as for outcome 1
Time Frame: Week 12
Population: ITT, subgroup of subjects that previously failed >=4 b/tsDMARD
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 30 | 34
Participants | 9 | 12
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.415, Cochran-Mantel-Haenszel; Risk Difference (RD) = -2.4, 95% CI 2-sided [-24.1 to 19.2]

ADVERSE EVENTS:
Time Frame: As collected from time of consent through March 10, 2025 (data cut date for Clinical Study Report). This period coverage an average duration of 803 days (2.2 years) for each subject.
Description: All AEs and SAEs were categorized by Co-PIs as related or not related to the implant procedure, the explant procedure, the Implant, the Charger, or stimulation.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/120
Serious Adverse Events (participants affected / at risk) | 22/122 | 29/120
Other Adverse Events (participants affected / at risk) | 74/122 | 79/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=122) | Control (N=120)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Related, Serious AEs from Implantation to Week 12
Incision site swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Related, Serious AEs from Implantation to Week 12
Pharyngeal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Related, Serious AEs from Implantation to Week 12
Vocal cord paresis (Nervous system disorders) | 1 (1) | 0 (0) — Related, Serious AEs from Implantation to Week 12
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs from Implantation to Week 12
Chest pain (General disorders and administration site conditions) | 0 (0) | 1 (1) — Unrelated, Serious AEs from Implantation to Week 12
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs from Implantation to Week 12
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs from Implantation to Week 12
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated, Serious AEs from Implantation to Week 12
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs from Implantation to Week 12
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated, Serious AEs from Implantation to Week 12
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs from Implantation to Week 12
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Benign abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Blood pressure increased (Investigations) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) — Unrelated, Serious AEs during Long-term Follow-up
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) — Unrelated, Serious AEs during Long-term Follow-up
Chest pain (General disorders and administration site conditions) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Device related infection (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Hypertension (Vascular disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Myocardial infarction (Cardiac disorders) | 1 (2) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Pain (General disorders and administration site conditions) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) — Unrelated, Serious AEs during Long-term Follow-up
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Retinal tear (Eye disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Rotator cuff syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Septic shock (Infections and infestations) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated, Serious AEs during Long-term Follow-up
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) — Unrelated, Serious AEs during Long-term Follow-up
Urosepsis (Infections and infestations) | 0 (0) | 1 (2) — Unrelated, Serious AEs during Long-term Follow-up
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=122) | Control (N=120)
Vocal cord paresis (Nervous system disorders) | 5 (5) | 6 (6) — Non-Serious Procedure or Implant Related AEs from Implant to Week 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) — Non-Serious Procedure or Implant Related AEs from Implant to Week 12
Medical device pain (General disorders and administration site conditions) | 4 (4) | 0 (0) — Non-Serious Stimulation Related AEs from Randomization to Week 12
COVID-19 (Infections and infestations) | 8 (8) | 6 (6) — Non-Serious Unrelated AEs from Implant to Week 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8) | 1 (1) — Non-Serious Unrelated AEs from Implant to Week 12
Sinusitis (Infections and infestations) | 3 (3) | 4 (4) — Non-Serious Unrelated AEs from Implant to Week 12
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) — Non-Serious Unrelated AEs from Implant to Week 12
Bronchitis (Infections and infestations) | 1 (1) | 4 (4) — Non-Serious Unrelated AEs from Implant to Week 12
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) — Non-Serious Unrelated AEs from Implant to Week 12
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) — Non-Serious Unrelated AEs from Implant to Week 12
Headache (Nervous system disorders) | 0 (0) | 4 (4) — Non-Serious Unrelated AEs from Implant to Week 12
COVID-19 (Infections and infestations) | 18 (21) | 23 (26) — Non-Serious Unrelated AEs During Long-term Follow-up
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (13) | 8 (8) — Non-Serious Unrelated AEs During Long-term Follow-up
Nasopharyngitis (Infections and infestations) | 10 (12) | 5 (5) — Non-Serious Unrelated AEs During Long-term Follow-up
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 2 (2) — Non-Serious Unrelated AEs During Long-term Follow-up
Sinusitis (Infections and infestations) | 9 (9) | 8 (10) — Non-Serious Unrelated AEs During Long-term Follow-up
Urinary tract infection (Infections and infestations) | 8 (12) | 10 (14) — Non-Serious Unrelated AEs During Long-term Follow-up
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (9) | 8 (8) — Non-Serious Unrelated AEs During Long-term Follow-up
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4) — Non-Serious Unrelated AEs During Long-term Follow-up
Carpal tunnel syndrome (Nervous system disorders) | 5 (5) | 2 (2) — Non-Serious Unrelated AEs During Long-term Follow-up
Bursitis (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) — Non-Serious Unrelated AEs During Long-term Follow-up
Nerve compression (Nervous system disorders) | 4 (4) | 0 (0) — Non-Serious Unrelated AEs During Long-term Follow-up
Hypertension (Vascular disorders) | 3 (4) | 4 (4) — Non-Serious Unrelated AEs During Long-term Follow-up
Influenza (Infections and infestations) | 3 (3) | 6 (6) — Non-Serious Unrelated AEs During Long-term Follow-up
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) — Non-Serious Unrelated AEs During Long-term Follow-up
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) — Non-Serious Unrelated AEs During Long-term Follow-up
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) — Non-Serious Unrelated AEs During Long-term Follow-up
Depression (Psychiatric disorders) | 1 (1) | 6 (6) — Non-Serious Unrelated AEs During Long-term Follow-up
Pain (General disorders and administration site conditions) | 1 (1) | 4 (5) — Non-Serious Unrelated AEs During Long-term Follow-up

LIMITATIONS AND CAVEATS:
A possible limitation was a 3-month controlled phase, which did not capture peak therapeutic response, known to evolve over longer periods for some patients based on prior experience with vagus nerve stimulation. This is likely influenced by modulation of innate neuroimmune pathways vs. inhibition of discrete inflammatory pathways, the mechanism of most pharmaceutical interventions. Nevertheless, consistency of outcomes across multiple visits thru Wk 48 supports durability of treatment effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT04539964/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT04539964/SAP_001.pdf